CLINICAL TRIAL: NCT05941468
Title: Using Augmented Reality Dental Care Training in Health Education on Periodontal Status, Blood Sugar Control and Quality of Life in Patients With Poorly Controlled Type 2 Diabetes
Brief Title: Using AR Dental Care Training System in HE on Periodontal Status, Blood Sugar Control and QoL in Patients With T2DM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kaohsiung Medical University Chung-Ho Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: KMUHIRB-F(II)-20230056
Record Dates: First submitted 2023-07-04; First posted 2023-07-12 (Actual); Last update posted 2023-07-12 (Actual); Status verified 2023-04

CONDITIONS: Diabetes Mellitus Type 2 With Periodontal Disease
Keywords: Augmented Reality; Periodontitis; Blood Sugar Control; Type 2 Diabetes
MeSH Terms: conditions — Periodontitis; Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- AR group (EG-A) (Experimental): Behavioral: AR intervention For the EG-A, the AR dental care training system will give to patients that 2 to 3 times tooth clean skill learning course (including Bass method of brushing and inter-dental toothbrush brushing technique) during non-surgical periodontal treatment period.
  Interventions: Device: AR Dental Care Training System
- AR-health consulting group (EG-B) (Experimental): Behavioral: AR intervention For the EG-B, the AR dental care training system will give to patients that 2 to 3 times tooth clean skill learning course (including Bass method of brushing and inter-dental toothbrush brushing technique) during non-surgical periodontal treatment period.
  The health counseling will also provide professional oral health related courses (including oral care for diabetes and periodontal disease, etc.)
  Interventions: Device: AR Dental Care Training System
- Control group (CG) (No Intervention): the control group(CG) only have standard oral hygiene education

INTERVENTIONS:
Device: AR Dental Care Training System — AR dental care training system is the first training system used in tooth clean skill learning (including Bass method of brushing and inter-dental toothbrush brushing technique) the world, it has been used to training elementary school children and dental hygiene student. And we are the first study to use this system to learn oral cleaning skill in hospital for patient with T2DM.
  Arms: AR group (EG-A); AR-health consulting group (EG-B)

SUMMARY:
The aim of this study was to evaluate the long-term effectiveness of an AR dental care training in health education on periodontal status, blood sugar control and quality of life in patients with poorly controlled type 2 diabetes. This randomized controlled trial included experimental group: AR group (EG-A), AR-health consulting group (EG-B) and control group (CG), respectively.

The EG-A and EG-B received AR dental care training intervention 2 to 3 times during non-surgical periodontal treatment.

Baseline and follow-up surveys were used to collect the data in periodontal index, blood sugar data, oral health knowledge, attitudes, behavior, oral health-related quality of life.

DETAILED DESCRIPTION:
A randomized experimental design was used. Patients with type 2 diabetes whose aged 35-65 years and HbA1c over 7% in the past six months were recruited through department of Endocrinology and Metabolism in Kaohsiung Medical University Hospital.

Each group was expected for 100 per group, patients will be randomized into each group. G*Power (version 3.1.9.4) was used for power analysis.

All patients will underwent periodontal examination at baseline and at 1-month, 3-month, 6-month and 1 year follow-ups.

Each patients will be diagnosed periodontal disease by dentist and have more than 12 functional teeth.

Each patients will completed the questionnaire at baseline and at 1-month, 3- month,6-month and 1 year follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Age 35 years old (inclusive) and above
* HbA1c over 7% in the past six months
* There are more than 12 functional teeth to ensure that the patient has enough teeth to evaluate the periodontal condition

Exclusion Criteria:

* Have received periodontal treatment within the previous 6 months
* Habits of smoking, drugs and betel nut chewing
* Taking antibiotics and osteoporosis bisphosphonates and other drugs regularly
* People with cognitive function or physical and mental disabilities
* Severely impaired diseases (for example: cancer, renal function or liver failure, etc.)

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-03-28 (Actual); Primary Completion 2024-03-27 (Estimated); Study Completion 2024-03-27 (Estimated)

PRIMARY OUTCOMES:
Gingival index (GI) | Change from Baseline GI at 1-month after intervention
  The gingiva inflammation status of 6 tooth was recorded using the gingiva index, as follows:
  0 = No inflammation.
  1. = Mild inflammation, slight change in color, slight edema, no bleeding on probing
  2. = Moderate inflammation, moderate glazing, redness, bleeding on probing
  3. = Severe inflammation, marked redness and hypertrophy, ulceration, tendency to spontaneous bleeding.
  For each patient, GI will measured by the teeth 12,16,24,32,36,44
Gingival index (GI) | Change from Baseline GI at 3-month after intervention
  The gingiva inflammation status of 6 tooth was recorded using the gingiva index, as follows:
  0 = No inflammation.
  1. = Mild inflammation, slight change in color, slight edema, no bleeding on probing
  2. = Moderate inflammation, moderate glazing, redness, bleeding on probing
  3. = Severe inflammation, marked redness and hypertrophy, ulceration, tendency to spontaneous bleeding.
  For each patient, GI will measured by the teeth 12,16,24,32,36,44
Gingival index (GI) | Change from Baseline GI at 6-month after intervention
  The gingiva inflammation status of 6 tooth was recorded using the gingiva index, as follows:
  0 = No inflammation.
  1. = Mild inflammation, slight change in color, slight edema, no bleeding on probing
  2. = Moderate inflammation, moderate glazing, redness, bleeding on probing
  3. = Severe inflammation, marked redness and hypertrophy, ulceration, tendency to spontaneous bleeding.
  For each patient, GI will measured by the teeth 12,16,24,32,36,44
Gingival index (GI) | Change from Baseline GI at 1 year after intervention
  The gingiva inflammation status of 6 tooth was recorded using the gingiva index, as follows:
  0 = No inflammation.
  1. = Mild inflammation, slight change in color, slight edema, no bleeding on probing
  2. = Moderate inflammation, moderate glazing, redness, bleeding on probing
  3. = Severe inflammation, marked redness and hypertrophy, ulceration, tendency to spontaneous bleeding.
  For each patient, GI will measured by the teeth 12,16,24,32,36,44
Plaque index (PI) | Change from Baseline PI at 1-month after intervention
  The plaque status of 6 tooth was recorded using the plaque index, as followes:
  0 = No plaque
  1. = Thin film of plaque, scraped with explorer
  2. = Moderate amount of plaque, visible with naked eyes
  3. = Abundance of soft matter within the gingival pocket and/or on the tooth and gingival margin.
  For each patient, PI will measured by the teeth 12,16,24,32,36,44
Plaque index (PI) | Change from Baseline PI at 3-month after intervention
  The plaque status of 6 tooth was recorded using the plaque index, as followes:
  0 = No plaque
  1. = Thin film of plaque, scraped with explorer
  2. = Moderate amount of plaque, visible with naked eyes
  3. = Abundance of soft matter within the gingival pocket and/or on the tooth and gingival margin.
  For each patient, PI will measured by the teeth 12,16,24,32,36,44
Plaque index (PI) | Change from Baseline PI at 6-month after intervention
  The plaque status of 6 tooth was recorded using the plaque index, as followes:
  0 = No plaque
  1. = Thin film of plaque, scraped with explorer
  2. = Moderate amount of plaque, visible with naked eyes
  3. = Abundance of soft matter within the gingival pocket and/or on the tooth and gingival margin.
  For each patient, PI will measured by the teeth 12,16,24,32,36,44
Plaque index (PI) | Change from Baseline PI at 1 year after intervention
  The plaque status of 6 tooth was recorded using the plaque index, as followes:
  0 = No plaque
  1. = Thin film of plaque, scraped with explorer
  2. = Moderate amount of plaque, visible with naked eyes
  3. = Abundance of soft matter within the gingival pocket and/or on the tooth and gingival margin.
  For each patient, PI will measured by the teeth 12,16,24,32,36,44
Probing Pocket Depth (PPD) | Change from Baseline PPD at 1-month after intervention
  Using periodontal probe to measure the depth from the bottom of the periodontal pocket to the gingival margin.
  For each patient, PPD will measured each teeth.
Probing Pocket Depth (PPD) | Change from Baseline PPD at 3-month after intervention
  Using periodontal probe to measure the depth from the bottom of the periodontal pocket to the gingival margin.
  For each patient, PPD will measured each teeth.
Probing Pocket Depth (PPD) | Change from Baseline PPD at 6-month after intervention
  Using periodontal probe to measure the depth from the bottom of the periodontal pocket to the gingival margin.
  For each patient, PPD will measured each teeth.
Probing Pocket Depth (PPD) | Change from Baseline PPD at 1 year after intervention
  Using periodontal probe to measure the depth from the bottom of the periodontal pocket to the gingival margin.
  For each patient, PPD will measured each teeth.
Clinical Attachment Loss(CAL) | Change from Baseline CAL at 1-month after intervention
  Using periodontal probe to measure the distance from the enamel-dentin junction to the bottom of the periodontal pocket.
  For each patient, CAL will measured each teeth.
Clinical Attachment Loss(CAL) | Change from Baseline CAL at 3-month after intervention
  Using periodontal probe to measure the distance from the enamel-dentin junction to the bottom of the periodontal pocket.
  For each patient, CAL will measured each teeth.
Clinical Attachment Loss(CAL) | Change from Baseline CAL at 6-month after intervention
  Using periodontal probe to measure the distance from the enamel-dentin junction to the bottom of the periodontal pocket.
  For each patient, CAL will measured each teeth.
Clinical Attachment Loss(CAL) | Change from Baseline CAL at 1 year after intervention
  Using periodontal probe to measure the distance from the enamel-dentin junction to the bottom of the periodontal pocket.
  For each patient, CAL will measured each teeth.
Plaque Control Record (PCR) | Change from Baseline PCR at 1-month after intervention
  The Plaque Control Record is a very simple percentage or score of the total amount of bacteria present in your mouth. A tooth has 6 surfaces at the gum line being; the lingual side (distal, middle, mesial) and buccal side (distal, middle, mesial).
  For each patient, PCR will measured each teeth.
Plaque Control Record (PCR) | Change from Baseline PCR at 3-month after intervention
  The Plaque Control Record is a very simple percentage or score of the total amount of bacteria present in your mouth. A tooth has 6 surfaces at the gum line being; the lingual side (distal, middle, mesial) and buccal side (distal, middle, mesial).
  For each patient, PCR will measured each teeth.
Plaque Control Record (PCR) | Change from Baseline PCR at 6-month after intervention
  The Plaque Control Record is a very simple percentage or score of the total amount of bacteria present in your mouth. A tooth has 6 surfaces at the gum line being; the lingual side (distal, middle, mesial) and buccal side (distal, middle, mesial).
  For each patient, PCR will measured each teeth.
Plaque Control Record (PCR) | Change from Baseline PCR at 1 year after intervention
  The Plaque Control Record is a very simple percentage or score of the total amount of bacteria present in your mouth. A tooth has 6 surfaces at the gum line being; the lingual side (distal, middle, mesial) and buccal side (distal, middle, mesial).
  For each patient, PCR will measured each teeth.

SECONDARY OUTCOMES:
Oral health knowledge | Change from Baseline at 1-month after intervention
  The oral health knowledge is a questionnaire scale. Total of 12 items ex. Are diabetic patients more likely to have periodontal disease? score range is 0 to 12, higher score means have the better the oral health knowledge.
Oral health knowledge | Change from Baseline at 3-month after intervention
  The oral health knowledge is a questionnaire scale. Total of 12 items ex. Are diabetic patients more likely to have periodontal disease? score range is 0 to 12, higher score means have the better the oral health knowledge.
Oral health knowledge | Change from Baseline at 6-month after intervention
  The oral health knowledge is a questionnaire scale. Total of 12 items ex. Are diabetic patients more likely to have periodontal disease? score range is 0 to 12, higher score means have the better the oral health knowledge.
Oral health knowledge | Change from Baseline at 1 year after intervention
  The oral health knowledge is a questionnaire scale. Total of 12 items ex. Are diabetic patients more likely to have periodontal disease? score range is 0 to 12, higher score means have the better the oral health knowledge.
Attitude toward oral health | Change from Baseline at 1-month after intervention
  The attitude toward oral health is a questionnaire scale. Total of 7 items ex. It's normal for older people to lose their teeth. score range is 7 to 35, higher score means have more positive attitude toward oral health.
Attitude toward oral health | Change from Baseline at 3-month after intervention
  The attitude toward oral health is a questionnaire scale. Total of 7 items ex. It's normal for older people to lose their teeth. score range is 7 to 35, higher score means have more positive attitude toward oral health.
Attitude toward oral health | Change from Baseline at 6-month after intervention
  The attitude toward oral health is a questionnaire scale. Total of 7 items ex. It's normal for older people to lose their teeth. score range is 7 to 35, higher score means have more positive attitude toward oral health.
Attitude toward oral health | Change from Baseline at 1 year after intervention
  The attitude toward oral health is a questionnaire scale. Total of 7 items ex. It's normal for older people to lose their teeth. score range is 7 to 35, higher score means have more positive attitude toward oral health.
Oral Health Related Quality of Life(OHRQoL) | Change from Baseline at 1-month after intervention
  The OHRQoL is a questionnaire scale. Total of 14 items 7 dimensions including functional limitation, physical discomfort, psychological discomfort, physical disability, psychological disability, social disability and handicaps score range is 0-56 points, the lower the score, the greater the OHRQoL
Oral Health Related Quality of Life(OHRQoL) | Change from Baseline at 3-month after intervention
  The OHRQoL is a questionnaire scale. Total of 14 items 7 dimensions including functional limitation, physical discomfort, psychological discomfort, physical disability, psychological disability, social disability and handicaps score range is 0-56 points, the lower the score, the greater the OHRQoL
Oral Health Related Quality of Life(OHRQoL) | Change from Baseline at 6-month after intervention
  The OHRQoL is a questionnaire scale. Total of 14 items 7 dimensions including functional limitation, physical discomfort, psychological discomfort, physical disability, psychological disability, social disability and handicaps score range is 0-56 points, the lower the score, the greater the OHRQoL
Oral Health Related Quality of Life(OHRQoL) | Change from Baseline at 1 year after intervention
  The OHRQoL is a questionnaire scale. Total of 14 items 7 dimensions including functional limitation, physical discomfort, psychological discomfort, physical disability, psychological disability, social disability and handicaps score range is 0-56 points, the lower the score, the greater the OHRQoL

CONTACTS AND LOCATIONS:
Overall Officials: HSIAO-LING HUANG, Dr.PH, Principal Investigator — Kaohsiung Medical University, College of Dental Medicine, Department of Oral Hygiene
Locations (1):
- Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City, Taiwan